CLINICAL TRIAL: NCT03881891
Title: Optimizing Acute Post-Operative Dental Pain Management Using New Health Information Technology
Acronym: AHRQPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A131587; U18HS026135 (AHRQ)
Record Dates: First submitted 2019-03-14; First posted 2019-03-20 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Pain, Postoperative; Complication, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow-app intervention arm (Experimental): This arm will comprise of patients who are prompted to complete the PROMIS pain intensity scale through text/Short Message Service(SMS) or email mobile device notifications at pre-defined time intervals on Days 1, 3, 5 and 7 post-operatively.
  Interventions: Behavioral: Follow-app intervention arm
- Standard care arm (No Intervention): This arm will comprise of patients who receive the usual care.

INTERVENTIONS:
Behavioral: Follow-app intervention arm — The intervention includes implementation and evaluation of the effectiveness of a mobile phone-based text messaging system (FollowApp.Care) to collect patients' assessments of their post-op symptoms (pain intensity) and to use that data to improve their quality of care (pain experience) in the dental office setting
  Arms: Follow-app intervention arm

SUMMARY:
The investigators seek to implement a dental patient reported outcomes system using mobile phone and text messaging to target the over-reliance on pre-emptively prescribed opioids by dental providers. If successful, this project will help dentists actively track and manage their patients' pain after hours and enhance the overall care experience.

DETAILED DESCRIPTION:
Pain has been deemed the fifth vital sign and many describe it as an adverse event. The adequate management of pain is the bane of the dental profession and its continuous assessment is crucial to minimizing patients' pain experiences. Due to the duration of action of most commonly-used local anesthetic agents, dental patients are unable to predict their pain following dental procedures until many hours later, when the participants have already returned home and dental offices are closed. This has led to an over-reliance on pre-emptively prescribed opioids by dental providers because the participants have no means to actively track their patients' pain after hours. Innovative mobile applications and connected health technologies that allow real-time tracking of patients' symptoms, functional status and quality of life, provide healthcare professionals with data that were previously unavailable, and have fostered patient engagement, shared decision-making and adherence to treatment plans. The investigators propose an innovative solution to optimize the quality of dental pain monitoring and management by implementing mobile phone technology to monitor patients' pain during the critical acute post-operative phase. The hypothesis is that by actively tracking these symptoms using mobile phones, the investigators modify analgesic prescriptions), thereby eliminating needless suffering, reducing the occurrence and/or severity of post-op complications, and enhancing the overall care experience. The investigators' ultimate goal is to achieve the quadruple aim: improve patient experience, improve patient outcomes, improve physician experience and reduce per capita costs. The investigators will test this hypothesis using a cluster-randomized experimental study design with: (1) an intervention arm where patients receive push notifications through text messages on their mobile phones (FollowApp.Care) at designated time intervals on Days 1, 3, 5 and 7; and (2) a control arm where patients receive the usual care. This project will be conducted at two dental institutions: Willamette Dental Group (WDG) and University of California San Francisco (UCSF). In Aim 1 the investigators will customize the design features of the existing FollowApp.Care at two dental institutions (Willamette Dental Group and University of California San Francisco) and assess its capacity to accurately capture patient-reported outcomes. In Aim 2 the investigators evaluate the impact of using FollowApp.Care on patient post-op experiences and oral health outcomes. And in Aim 3, the investigators evaluate provider acceptance of FollowApp.Care and its impact on provider performance. By collecting patient reported outcomes in a timely and usable way, the investigators expect to help dentists enhance their practice performance and reduce the burden of unnecessary opioid prescriptions on society.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone periodontal procedures.
* Patients who have undergone endodontic procedures.
* Patients who have undergone oral surgery procedures.

Exclusion Criteria:

* 3rd year pre-doctoral students
* 4th year pre-doctoral students
* dental hygiene students

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1525 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity in the intervention arm, measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v.1.0 survey instrument | On day 1 post procedure for each patient.
  Evaluate the pain intensity on Day 1 following completion of the specified dental procedures. Raw scores for the pain intensity construct are determined by summing each of the individual scores from the three questions for each participant. The raw scores are then standardized using a T-score, which ranges from 0 to 100 with a mean of 50 and standard deviation of 10. Scores closer to 100 indicate high pain intensities and scores closer to 0 indicate lower pain intensities.
Pain intensity in the intervention arm, measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v.1.0 survey instrument | On day 3 post procedure for each patient.
  Evaluate the pain intensity on Day 3 following completion of the specified dental procedures. Raw scores for the pain intensity construct are determined by summing each of the individual scores from the three questions for each participant. The raw scores are then standardized using a T-score, which ranges from 0 to 100 with a mean of 50 and standard deviation of 10. Scores closer to 100 indicate high pain intensities and scores closer to 0 indicate lower pain intensities.
Pain intensity in the intervention arm, measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v.1.0 survey instrument | On day 5 post procedure for each patient.
  Evaluate the pain intensity on Day 5 following completion of the specified dental procedures. Raw scores for the pain intensity construct are determined by summing each of the individual scores from the three questions for each participant. The raw scores are then standardized using a T-score, which ranges from 0 to 100 with a mean of 50 and standard deviation of 10. Scores closer to 100 indicate high pain intensities and scores closer to 0 indicate lower pain intensities.
Pain intensity in the intervention arm, measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v.1.0 survey instrument | On day 7 post procedure for each patient.
  Evaluate the pain intensity on Day 7 following completion of the specified dental procedures. Raw scores for the pain intensity construct are determined by summing each of the individual scores from the three questions for each participant. The raw scores are then standardized using a T-score, which ranges from 0 to 100 with a mean of 50 and standard deviation of 10. Scores closer to 100 indicate high pain intensities and scores closer to 0 indicate lower pain intensities.
Pain experience in both arms, measured using the American Pain Society, the Patient Outcome Questionnaire (APS-POQ-R) questionnaire. | The pain experience outcome will be measured 7 days post procedure.
  Assess patients' 7-day post-op pain experiences. The dependent variables for our analysis will be derived from the questions: "How often were you in severe pain in the first 7 days?" A score of zero signifies that the respondent was "never in severe pain" while a score of 100 means the patient was "always in severe pain"; and 2b) "How satisfied you are with the results of your pain treatment following your dental procedure?" The patient satisfaction outcome scale ranges from 0 to 10 with low scores representing low satisfaction and higher scores representing higher satisfaction.
Provider Acceptance of FollowApp.Care | 2nd Quarter Year 3
  The investigators will administer the 26-item Technology Acceptance Model (TAM2) Questionnaire to providers in the intervention group pre- and post-implementation, to assess their perceived usefulness and perceived ease of use of FollowApp.Care as predictors of their usage behavior. The control group will also be invited to complete the TAM2 questionnaire post-implementation only, to assess their
  acceptance of FollowApp.Care if it is made available to them.

SECONDARY OUTCOMES:
Unscheduled/emergency visits during the study period; | through study completion, an average of 3 years
  This measure will be compiled on a monthly basis through chart review. At the patient level, the distribution of emergency/unscheduled follow-up visits (frequency and mean) will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Elsbeth Kalenderian, DDS, PhD, Principal Investigator — University of California, San Francisco; Muhammad F Walji, PhD, Principal Investigator — UT Houston
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Willamette Dental Group & Skourtes Institute, Hillsboro, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tokede B, Yansane A, Ibarra-Noriega A, Mullins J, Simmons K, Skourtes N, Mehta U, Tungare S, Holmes D, White J, Walji M, Kalenderian E. Evaluating the Impact of an mHealth Platform for Managing Acute Postoperative Dental Pain: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Oct 20;11:e49677. doi: 10.2196/49677. PMID 37933185

DOCUMENTS (4):
  • Informed Consent Form: Patient Control (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03881891/ICF_000.pdf
  • Informed Consent Form: Patient Intervention (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03881891/ICF_001.pdf
  • Informed Consent Form: Provider Control (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03881891/ICF_002.pdf
  • Informed Consent Form: Povider Intervention (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03881891/ICF_003.pdf